CLINICAL TRIAL: NCT02593422
Title: Writing About Experiences With Ovarian Cancer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 728101-3
Record Dates: First submitted 2015-10-26; First posted 2015-11-02 (Estimated); Last update posted 2022-05-23 (Actual); Status verified 2022-05

CONDITIONS: Ovarian Cancer
Keywords: ovarian cancer; expressive writing; writing interventions; psychosocial support
MeSH Terms: conditions — Ovarian Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- Expressive Writing (Experimental): Writing about ovarian cancer: Participants will be asked to write about their deepest thoughts and emotions about their experience with ovarian cancer
  Interventions: Behavioral: Expressive Writing
- Fact Writing (Control) (Active Comparator): Writing about ovarian cancer: Participants will be asked to write about the facts of their experience with ovarian cancer
  Interventions: Behavioral: Fact Writing (Control)

INTERVENTIONS:
Behavioral: Expressive Writing — Participants will be asked to write about their deepest thoughts and emotions about their experience with ovarian cancer
  Arms: Expressive Writing
Behavioral: Fact Writing (Control) — Participants will be asked to write about the facts of their experience with ovarian cancer
  Arms: Fact Writing (Control)

SUMMARY:
This online study aims to understand whether writing about one's experiences with ovarian cancer may be beneficial for psychological and physical wellbeing in women with a history of ovarian cancer. Investigators are also interested in studying how certain individual characteristics may impact the effectiveness of writing. Participants will be asked to complete an initial survey (15 min), followed by writing about their experiences with ovarian cancer on four occasions (20 - 25 min each), over the course of two weeks. A final survey (10 min) will be completed one month afterwards.

DETAILED DESCRIPTION:
The purpose of this randomized controlled experiment is to examine the effects of writing about experiences with ovarian cancer on psychological and physical outcomes in English-speaking women with a history of ovarian cancer. It will also examine how certain individual characteristics may impact the effectiveness of the writing interventions for different women. After completing an initial survey, women will be asked to write about their experiences with ovarian cancer on 4 separate occasions of 20-25 min each in the course of 2 weeks. A final survey will be completed one month after the last writing session. The entire study will be conducted online.

ELIGIBILITY:
Inclusion Criteria:

* Women with a history of ovarian cancer (any stage)
* At least 18 years old
* English-speaking/Can comfortably read and write in English
* Able to provide informed consent
* Internet access
* Valid email address
* Any region/country

Exclusion Criteria:

* Minors (younger than 18)
* Lack of English proficiency
* Inability to provide informed consent
* Male

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 73 (Actual)
Dates: Start 2015-04; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Change in Psychological Functioning (Wellbeing/Distress) | 6 - 9 weeks, with timely completion of writing: Initial survey (day 1), after 2nd writing task (week 1), after 4th writing task (week 2), and one month after last writing task (week 6)
  Various aspects of social, emotional and functional wellbeing will be assessed using the Functional Assessment of Cancer-Ovarian measure (FACT-O, Version 4, Basen-Engquist et al, 2001). Distress about ovarian cancer will be assessed using the Impact of Event Scale (IES, Horowitz, Wilner & Alvarez, 1979).

SECONDARY OUTCOMES:
Change in Physical Wellbeing | 6 - 9 weeks, with timely completion of writing: Initial survey (day 1), after 2nd writing task (week 1), after 4th writing task (week 2), and one month after last writing task (week 6)
  Physical symptoms and concerns specific to ovarian cancer will be assessed using Functional Assessment of Cancer - Ovarian (FACT-O, Version 4, Basen-Engquist et al, 2001).
Changes in affect before and after writing about ovarian cancer | Prior to and after each of 4 writing tasks (weeks 1 - 2)
  Positive and negative affect will be assessed using the Positive and Negative Affect Scale (PANAS, Watson, Clark & Tellegen, 1988).

CONTACTS AND LOCATIONS:
Overall Officials: Mary Ann Hoffman, Ph.D., Study Chair — University of Maryland, College Park
Locations (1):
- University of Maryland, College Park, College Park, Maryland, United States

REFERENCES:
- [Background] Merz EL, Fox RS, Malcarne VL. Expressive writing interventions in cancer patients: a systematic review. Health Psychol Rev. 2014;8(3):339-61. doi: 10.1080/17437199.2014.882007. Epub 2014 Feb 18. PMID 25053218
- [Background] Frattaroli J. Experimental disclosure and its moderators: a meta-analysis. Psychol Bull. 2006 Nov;132(6):823-65. doi: 10.1037/0033-2909.132.6.823. PMID 17073523